CLINICAL TRIAL: NCT01285778
Title: Phase 2 Trial to Assess the Efficacy and Safety of Chemoradiation With 5-fluorouracil, Mytomicin C and Panitumumab as a Treatment for Anal Squamous Cell Carcinoma
Brief Title: Vectibix for the Treatment of Anal Cancer
Acronym: VITAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Collaborators: Amgen (Industry); Trial Form Support S.L. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD-0902
Record Dates: First submitted 2011-01-20; First posted 2011-01-28 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Anal Squamous Cell Carcinoma
Keywords: Anal squamous cell carcinoma; panitumumab; chemoradiation; anal cancer; GEMCAD-09-02
MeSH Terms: conditions — Anus Neoplasms | interventions — Panitumumab; Fluorouracil; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab, mytomicin C, 5-FU, radiation (Experimental)
  Interventions: Drug: panitumumab, mytomicin C, 5-FU, radiation

INTERVENTIONS:
Drug: panitumumab, mytomicin C, 5-FU, radiation — Radiation therapy will be administered concurrent with chemotherapy and Panitumumab treatment. It will start the day 1 of the systemic treatment. That is, the first day of radiation therapy will be the day of the administration of the first dose of Panitumumab and Mitomycin C, as well as the first day of the first 96-hours course of 5-FU continuous infusion. On day 1, drugs and radiation will be administered in the following order:
  * First, Panitumumab. Panitumumab will be administered by IV infusion on day 1, and every 2 weeks during 8 weeks
  * Then Mitomycin C, 10mg/m2 on days 1 and 29
  * Then start the 5-FU continuous infusion, 1000mg/m2 on days 1-4 and 29-32
  * Finally, no less than 2 hours after the start of the 5-FU infusion, first dose of radiation therapy.
  Other Names: Vectibix

SUMMARY:
Chemoradiation with 5-FU and Mitomycin C is the standard treatment in anal canal SCC. Panitumumab has shown efficacy in other tumors and anti-EGFR treatment has shown clinical activity in a single report of a refractory anal canal SCC patient. Based on this background, we propose to conduct a phase II study to investigate the efficacy and toxicity of radiotherapy with the association:

* 5-FU 1000mg/m2 on days 1-4 and 29-32
* Mitomycin C 10mg/m2 on days 1 and 29
* Panitumumab 6 mg/kg on day 1, then every 2 weeks for 8 weeks

DETAILED DESCRIPTION:
In the 1980s, the treatment of choice for anal cancer was abdominal-perineal amputation, which included the removal of the anus, rectum and lymphatic drainage areas and a permanent colostomy. With this treatment, 5-year survival rates were 40-70%. In the following years, however, it was shown that anal cancer was a tumor that was sensitive to chemotherapy and radiation, so surgery was not the first choice and was only reserved for resistant cases or relapses. Concomitant chemo and radiotherapy based on the Mitomycin C - 5-FU regimen is currently the standard treatment for localized (except T1N0) and locally advanced cases. This statement is supported by two randomized studies that showed that the administration of chemoradiation with Mitomycin C - 5FU was better than radiation in monotherapy. The trial conducted by the United Kingdom Coordinating Committee on Cancer Research (UKCCCR) randomized 585 patients to receive radiotherapy (45 Gy in 4-5 weeks) or the same radiotherapy regimen coupled with 5-FU (1000 mg/m2 x 4 days or 750 mg/m2 x 5 days), for the first and last week of radiotherapy and Mitomycin C 12 mg/m2 on day 1. The 3-year local failure rate was 39% in the combined arm versus 61% with radiotherapy alone. There were no differences in the 3-year overall survival rate. On the other hand, in the study conducted by EORTC, 110 patients were distributed to receive radiotherapy (45 Gy in 5 weeks, with an overimpression of 15 Gy in the patients with CR and 20 Gy if PR) or radiotherapy plus 5-FU (750 mg/m2 days 1-5 and 29-33) associated to Mitomycin C (15 mg/m2 on day 1). The CR rate was significantly greater in the group treated with chemoradiation (80% vs. 54%). After 5 years of follow-up, there was still an 18% increase in the local control rate in favor of the group treated with chemoradiation.

More recently, the results of a phase II CALGB trial, suggests that the administration of induction treatment with two cycles of cisplatin-5FU (cisplatin 100 mg/m2 on days 1 and 29 and 5FU 1000 mg/m2 days 1-4 and 29-32) followed by chemoradiotherapy with 5-FU and Mitomycin C was very promising, especially in patients with a poor prognosis, with 50% of patients remaining colostomy and disease-free at 48 months. However, in a randomized study by the RTOG group, which included 682 patients, this strategy was compared with the classic concomitant chemoradiation with 5-FU (1000 mg/m2 days 1-4 and 29-32) and Mitomycin C (10 mg/m2 days 1 and 29). No differences in survival were found, but it was also detected that the colostomy rate was greater in the patients treated with the regimen containing Cisplatin (HR, 1.68; 95% CI, 1.07-2.65; P=.02). The authors concluded that induction with cisplatin was not superior to the traditional administration of 5FU-Mitomycin C with RT.

Epidermoid anal cancer is a tumor that often expresses the EGFR receptor. In an initial study with 21 cases, it was reported that there was EGFR expression in all the biopsies. In another study with 38 cases, it was found that 55% of the tumors expressed EGFR. No study has been published, however, which has investigated the efficacy of Panitumumab in this tumor. There is only one report of a refractory case in which cetuximab was administered together with CPT-11 with an excellent response.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman ≥ 18 years
* Competent to comprehend, sign, and date an IEC-approved informed consent form
* Histologically or cytologically-confirmed anal canal SCC
* T status 2-4 and any N status (pelvic or inguinal) radiologically defined by MRI
* De novo diagnosis of anal canal SCC not previously treated
* ECOG performance status of 0, 1 or 2
* If a subject has prior history of cancer other than anal canal SCC, non-melanoma skin carcinoma, or in situ cervical carcinoma, then the subject should neither have received any treatment nor have shown any signs of active disease within the previous 5 years
* Adequate bone marrow function: neutrophils≥1.5 x109/ L; platelets≥100 x109/ L; hemoglobin≥ 9 g/ dL
* Hepatic function as follows: total bilirubin count ≤ 1.5 x ULN; ALT and AST ≤ 2.5 x ULN
* Calculated creatinine clearance or 24 hour creatinine clearance ≥ 50 mL/ min
* Magnesium≥ lower limit of normal

Exclusion Criteria:

* Metastatic anal canal SCC
* HIV infection (except patients with an undetectable viral load and CD4 cells count >400/mL which are eligible for the study)
* Known hypersensitivity to any of the study drugs
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications
* Patients they have received prior systemic therapy or radiotherapy for the treatment of SCC anal carcinoma.
* Prior malignant tumor in the last 5 years, except a history of non-melanoma skin carcinoma, or in situ cervical carcinoma.
* Clinically significant cardiovascular disease, for example myocardial infarction (< 6 months before treatment start), unstable angina, congestive heart failure, arrhythmia requiring medication, or uncontrolled hypertension
* Known positive test for, hepatitis C virus, chronic active hepatitis B infection
* Any kind of disorder that compromises the ability of the subject to give written informed consent and/or comply with the study procedures
* Any investigational agent within 30 days before enrolment
* Subject who is pregnant or breast feeding
* Surgery (excluding diagnostic biopsy or central venous catheter placement) and/or radiotherapy within 28 days prior to inclusion in the study.
* Woman or man of childbearing potential not consenting to use adequate contraceptive precautions i.e. double barrier contraceptive methods (eg diaphragm plus condom), or abstinence during the course of the study and for 6 months after the last study drug administration for women, and 3 month for men
* Psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Three-year disease-free survival rate | 3 years
  To estimate the three-year disease-free survival rate in patients treated with 5-FU, mytomicin C and Panitumumab concurrently with radiation therapy as treatment for anal squamous cell carcinoma

SECONDARY OUTCOMES:
Disease free survival rate | 3 years
  To assess disease free survival in patients treated with 5-FU, Mytomicin C and Panitumumab concurrently with radiation therapy as treatment for anal squamous cell carcinoma.
Three-year free local-regional failure rate | 3 years
  To assess three-year free local-regional failure rate in patients treated with 5-FU, Mytomicin C and Panitumumab concurrently with radiation therapy as treatment for anal squamous cell carcinoma.
Overall survival | 3 years
  To assess overall survival in patients treated with 5-FU, Mytomicin C and Panitumumab concurrently with radiation therapy as treatment for anal squamous cell carcinoma.
Colostomy-free survival rate | 2 years
  To assess two-year colostomy-free survival rate in patients treated with 5-FU, Mytomicin C and Panitumumab concurrently with radiation therapy as treatment for anal squamous cell carcinoma.
Complete response rate | 3 years
  To assess complete response rate in patients treated with 5-FU, Mytomicin C and Panitumumab concurrently with radiation therapy as treatment for anal squamous cell carcinoma.
Safety profile | 3 years
  * Incidence of adverse events (including all serious, grade 3, grade 4, and treatment related events)
  * Changes in laboratory values.
Predictive potential of different biomarkers | 3 years
  * To investigate the predictive potential of different biomarkers involved in different pathways on efficacy and/or safety endpoints:
    1. EGFR pathway
    2. DNA reparation mechanisms and apoptosis control
    3. Oxidative stress control mechanism
    4. Resistance mechanisms to alkylants (mitomycin C) and antimetabolits (5-FU)
  * To describe the presence of HPV infection, isotype study and impact of the status on efficacy and/or safety.
  * To evaluate the role of magnetic resonance imaging (MRI) in the determination of therapeutic efficacy and follow-up of these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Feliu, MD, Study Director — Hospital Universitario La Paz; Vicente Alonso, MD, Principal Investigator — Hospital Miguel Servet; Jaume Capdevila, MD, Principal Investigator — Hospital Universitario Vall Hebron; Ruth Vera, MD, Principal Investigator — Hospital de Navarra; Miriam Lopez, MD, Principal Investigator — Hospital Infanta Sofia; Carmen Castañon, MD, Principal Investigator — Hospital Virgen Blanca (León); Carlos Fernández-Martos, MD, Principal Investigator — Instituto Valenciano de Oncología; Clara Montagut, MD, Principal Investigator — Hospital del Mar; Carlos García Girón, MD, Principal Investigator — Hospital General Yagüe (Burgos); Ana León, MD, Principal Investigator — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz; Marta Martín, MD, Principal Investigator — Hospital de la Santa Creu i Sant Pau de Barcelona; Juan Carlos Méndez, MD, Principal Investigator — Centro Oncológico de Galicia; Rocío García Carbonero, MD, Principal Investigator — Hospital Universitario Virgen del Rocío (Sevilla); Jordi Remon, MD, Principal Investigator — Hospital de Mataró; Fernando Rivera, MD, Principal Investigator — Hospital Universitario Marqués de Valdecilla (Santander); Laura Cerezo, MD, Principal Investigator — Hospital Universitario La Princesa (Madrid); Pilar García-Alfonso, MD, Principal Investigator — Hospital Universitario Gregorio Marañón (Madrid); Emilio Fonseca, MD, Principal Investigator — University of Salamanca; Aleydis Pisa, MD, Principal Investigator — Corporació Sanitaria Parc Taulí (Sabadell, Barcelona); Mónica Caro, MD, Principal Investigator — Institut Català d´Oncologia. Hospital Germans Trias i Pujol (Badalona); José María Vicent, MD, Principal Investigator — Hospital de Manises, Valencia; Isabel Sevilla, MD, Principal Investigator — Hospital Universitario Virgen de la Victoria (Málaga); Joan Maurel, MD, Principal Investigator — Hospital Clinic of Barcelona; I Guasch, MD, Principal Investigator — Hospital Sant Joan de Deu; Jesus Garcia-Foncillas, MD, Principal Investigator — Clinica Universidad de Navarra; Antonio Arrivi, MD, Principal Investigator — Hospital Son Llatzer
Locations (20):
- Spain (20):
  - Hospital Universitario Germans Trias i Pujol. Institut Català Oncologia, Badalona, Barcelona
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Centro Oncológico de Galicia, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall Hebron, Barcelona
  - Hospital Clínic i Provincial, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Virgen Blanca, León
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital General de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza